CLINICAL TRIAL: NCT00719173
Title: Evaluating the Effect of Aprepitant on Cyclophosphamide Pharmacokinetics
Brief Title: Effect of Aprepitant on Cyclophosphamide Pharmacokinetics in Patients With Breast Cancer
Acronym: NRR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCCC 0514; P30CA016086 (NIH); CDR0000600836 (Other: PDQ number); UNC-05-2917; UNC-GCRC-2411-ORC
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2024-11-04 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer; Nausea and Vomiting
Keywords: nausea and vomiting; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Nausea; Vomiting | interventions — Aprepitant; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive aprepitant 125 mg orally once daily on day 1 and 80 mg orally once daily on days 2 and 3. Beginning 1 hour after receiving aprepitant, patients receive an infusion of cyclophosphamide on day 1. During course 2, patients crossover and receive treatment as in arm II.
  Interventions: Drug: aprepitant; Drug: cyclophosphamide; Other: placebo
- Arm II (Experimental): Patients receive a placebo 125 mg orally once daily on day 1 and 80 mg orally once daily on days 2 and 3. Beginning 1 hour after receiving the placebo, patients will receive an infusion of cyclophosphamide infusion on day 1. During course 2, patients crossover and receive treatment as in arm I.
  Interventions: Drug: aprepitant; Drug: cyclophosphamide; Other: placebo

INTERVENTIONS:
Drug: aprepitant — Given orally
Drug: cyclophosphamide — Given IV
Other: placebo — Given orally

SUMMARY:
RATIONALE: Antiemetic drugs, such as aprepitant, may help lessen or prevent nausea and vomiting in patients undergoing chemotherapy.

PURPOSE: This randomized clinical trial is studying aprepitant to see how well it works compared to placebo in preventing nausea and vomiting in patients undergoing chemotherapy for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the effect of aprepitant on cyclophosphamide and 4-hydroxycyclophosphamide pharmacokinetics as measured by plasma AUC in patients with breast cancer.

Secondary

* To evaluate total control of nausea and vomiting, as defined by no vomiting episodes and no use of rescue medication, 72 hours after courses 1 and 2 of chemotherapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive aprepitant 125 mg orally once daily on day 1 and 80 mg orally once daily on days 2 and 3. Beginning 1 hour after receiving aprepitant, patients receive an infusion of cyclophosphamide on day 1. During course 2, patients crossover and receive treatment (placebo) as in arm II.
* Arm II: Patients receive a placebo 125 mg orally once daily on day 1 and 80 mg orally once daily on days 2 and 3. Beginning 1 hour after receiving the placebo, patients will receive an infusion of cyclophosphamide infusion on day 1. During course 2, patients crossover and receive treatment (aprepitant) as in arm I.

Patients complete a diary documenting nausea and vomiting on days 1, 2, and 3 of both courses. Patients also complete The Functional Living Index-Emesis (FLIE) questionnaire documenting compliance, rescue antiemetic therapy, and any adverse effects and record them in the diary for each course. Information in the patient's diary is obtained by the coordinator via telephone on day 4 of each course.

Patients undergo blood sample collection periodically for pharmacokinetic studies via high performance liquid chromatography.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* Planning to receive cyclophosphamide 600 mg/m²-1,000 mg/m² IV infusion

  * No cyclophosphamide dose change between courses 1 and 2

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 2 months
* ANC ≥ 1,500/μL
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 9.0 g/dL
* Serum creatinine ≤ 1.5 mg/dL
* AST/ALT ≤ 2 times upper limit of normal
* Not pregnant or nursing
* No contraindication to aprepitant

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent medications that are CYP3A4 substrates, inhibitors, and/or inducers, with the exception of the dexamethasone contained as part of the standard antiemetic regimen

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Effect of aprepitant on cyclophosphamide and 4-hydroxycyclophosphamide pharmacokinetics as measured by plasma AUC | 05/2005 to 10/2010
  Cyclophosphamide, 4-OH cyclophosphamide, and DCE PK with and without aprepitant

CONTACTS AND LOCATIONS:
Overall Officials: Christine M. Walko, PharmD, BCOP, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Walko CM, Combest AJ, Spasojevic I, Yu AY, Bhushan S, Hull JH, Hoskins J, Armstrong D, Carey L, Collicio F, Dees EC. The effect of aprepitant and race on the pharmacokinetics of cyclophosphamide in breast cancer patients. Cancer Chemother Pharmacol. 2012 May;69(5):1189-96. doi: 10.1007/s00280-011-1815-5. Epub 2012 Jan 15. PMID 22245954
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials